CLINICAL TRIAL: NCT03960060
Title: Evaluation of CAR (Chimeric Antigen Receptor) Modified Autologous T Cell CCT301-59 in Patients With Recurrent or Refractory Solid Tumors on the Basis of Safety, Tolerability and Anti-tumor Activity Study.
Brief Title: A Study of CCT301-59 CAR T Therapy in Adult Subjects With Recurrent or Refractory Solid Tumors
Acronym: CAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of study strategy
Sponsor: Shanghai PerHum Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT301-59-mST01
Record Dates: First submitted 2019-05-08; First posted 2019-05-22 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor; Soft Tissue Sarcoma; Gastric Cancer; Pancreatic Cancer; Bladder Cancer
MeSH Terms: conditions — Sarcoma; Stomach Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCT301-59 (Experimental): The safety and preliminary therapeutic efficacy of CCT301-59 will be evaluated for subjects with ROR2 positive biopsy in a standard 3+3 dose escalation rule. Three dose levels of CAR T will be administered in this study: 1x10^6, 3x10^6, 1x10^7 CCT301-59 CAR positive T cells/kg weight, intravenous infusion.
  Interventions: Biological: CCT301-59

INTERVENTIONS:
Biological: CCT301-59 — Collect blood from the patients and isolate peripheral blood mononuclear cells for the production of CCT301-59. Subjects will receive the conditioning chemotherapy regimen of cyclophosphamide and fludarabine for lymphodepletion during the production of CCT301-59 and then subjects will receive one dose of CCT301-59 via intravenous injection.

SUMMARY:
This clinical study is to investigate the safety and tolerability of CAR modified autologous T cells (CCT301-59) in subjects with recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
This is a single arm, open label, dose escalation clinical study to evaluate the safety and preliminary therapeutic efficacy of CCT301-59 T cells in adult subjects with relapsed and refractory stage IV metastatic solid tumors (soft tissue sarcoma, gastric cancer, pancreatic cancer, bladder cancer etc.).

The subjects with ROR2 (receptor tyrosine kinase-like orphan receptor 2) positive biopsy will receive CCT301-59.

According to the 3+3 rules during the dose escalation stage to receive CCT301-59 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary to participate in the clinical study, subjects and their family members agree to sign the informed consent form and follow all trial procedures.
2. Male or female subjects 18-70 years of age.
3. Subjects are diagnosed as recurrent or refractory solid tumors (soft tissue sarcoma, gastric cancer, pancreatic cancer and bladder cancer) with identified unresectable advanced or metastatic tumors by radiology and histology or cytology, progression after the first line or above treatment, or intolerance to standard treatment.
4. At least one measurable lesion in accordance with RECIST 1.1, the long diameter of non-lymph node lesions ≥10mm (millimeter) according to CT (computerized tomography) scan-sectional image, or the short diameter of lymph node lesions ≥15mm; the longest axis of the measurable lesion ≥10 mm in CT scan (CT scan layer ≤ 5mm); FDG PET (fluorodeoxyglucose -positron emission tomography) of the measurable lesion > 3 SUV (standardized uptake values).
5. Subjects with ROR2 positive tumor tissue: the percentage of ROR2 positive staining cells in tumor cells detected by immunohistochemistry or RNA (Ribonucleic acid) in situ hybridization is ≥ 50%. The samples could be used within one year , otherwise the sample will be re-collected for biopsy.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score is 0 to 1.
7. Expected survival will be ≥ 12 weeks.
8. The organ and hematopoietic functions must meet the following requirements:

   * Hemoglobin (HGB)≥90 g/L (gram per litre), no blood transfusion within two weeks;
   * White blood cell count (WBC) ≥ 2.5×10^9/L;
   * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L;
   * Platelet count (PLT) ≥ 80×10^9/L;
   * Total bilirubin (TBIL) ≤ 3.0ng/dL or ≤ 5 ULN (Upper Limit of Normal);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; AST and ALT≤ 5×ULN in case the abnormal hepatic function is caused by hepatocellular carcinoma or liver metastasis from other tumors;
   * Serum creatinine (Cr) ≤ 1.5×ULN; or creatinine clearance (CrCl) ≥ 50 mL/min (milliliter per minute);
9. Prothrombin time (PT): INR (International Normalized Ratio) <1.7 or prolonged, PT prolonged < 4 seconds from normal level;
10. Normal neurologic evaluation;
11. Sufficient venous access for venous intravenous blood collection and infusion, no other contraindications for blood cell separation;
12. Able to receive treatment and follow-up, including the treatment at the enrolled site;
13. Female subjects of childbearing age must take acceptable measures to minimize the possibility of pregnancy during the trial. The serum or urine pregnancy test must be negative prior to pre-treatment for female subjects of childbearing age;

Exclusion Criteria:

1. Pregnant or breastfeeding female subjects;
2. Active infection of hepatitis B, or active hepatitis C;
3. Infection with HIV/AIDS (Human Immunodeficiency Virus / Acquired Immunodeficiency Syndrome);
4. Other active infection with clinical significance;
5. Previous diseases or concurrent diseases:

   Subjects diagnosed as serious autoimmune disease in long-term (over two months) requirement of systemic immunosuppressant (steroid), or as immune mediated symptomatic diseases including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune vasculitis (e.g., Wegener's granulomatosis);
6. Subjects with previous diagnosis as motor neuron disease;
7. Subjects with previous disease of toxic epidermal necrolysis;
8. Having any mental disorder that may affect the understanding of informed consent and relevant questionnaires, including dementia, altered mental status;
9. Having serious uncontrollable disease judged in the study that may affect the subjects receiving the study treatment;
10. Subjects with other active malignant tumors in the past five years including basal or squamous cell skin cancer, superficial bladder cancer or in situ breast cancer who have been completely cured, and without any follow-up treatment are not included;
11. Current using of systemic steroid or steroid inhalant;
12. Have used of immunotherapy treatment in the past three months or PD-1 (Programmed cell death protein 1) antibody, PD-L1 (Programmed death-ligand 1) antibody, PD-L2 antibody, CD137 (tumor necrosis factor receptor superfamily member 9, 4-1BB) antibody or CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) antibody, or cell therapy.
13. Allergy to immunotherapy or relevant medications;
14. Meningeal metastasis or central nervous system metastasis in the last 6 months, with obvious underlying diseases of the central nervous system, and leaving obvious symptoms;
15. Subjects with NYHA (New York Heart Association) heart failure grade ≥ 2 or uncontrollable hypertension by standard treatment and requiring special treatment, or with history of myocarditis, or occurrence of myocardial infarction within one year;
16. Previous organ transplantation or be ready for organ transplantation;
17. Pancreatic cancer with pancreatitis;
18. Active bleeding;
19. Subjects with pleural effusion or abdominal effusion that require clinical treatment or intervention;
20. Being judged by investigators as inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety of CCT301-59 CAR T cell therapy | Up to 52 weeks
  To observe the safety of CCT301-59 CAR positive T cells in subjects using Common Toxicity Criteria for Adverse effects (CTCAE) version 5.0.
Efficacy of CCT301-59 CAR T cell therapy | Up to 52 weeks
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Kinetics of CAR T cells | Up to 52 weeks
  The level of CAR T cells in the peripheral blood and persistence of CAR T cells in patients will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Zhou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China